CLINICAL TRIAL: NCT05189821
Title: RFA Treatment for Papillary Thyroid Microcarcinoma Cohort
Brief Title: RFA Treatment for Papillary Thyroid Microcarcinoma
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jennifer Kuo, Associate Professor, Columbia University
Other Study IDs: AAAT6770
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Papillary Thyroid Microcarcinoma
Keywords: Radiofrequency Ablation
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Ultrasound guided radiofrequency ablation

SUMMARY:
Thyroid surgery has always been the mainstay of treatment for thyroid cancer. Thyroid surgery carries a low risk of complications that include recurrent or superior laryngeal nerve injury leading to voice changes, hypoparathyroidism, hypothyroidism with need for thyroid hormone supplementation, and unsightly scarring. Although many patients with thyroid cancer find these risks acceptable, these risks are sometimes less acceptable to patients with benign disease. In an era when the medical field is treating thyroid diseases less aggressively, there is a pressing need to identify approaches to treat indolent malignant disease less invasively.

The purpose of this observational study is to evaluate the efficacy and safety of Radiofrequency Ablation (RFA) for treatment of Papillary Thyroid Microcarcinoma (PTMC) in patients that have already agreed to RFA procedure based on treating physician recommendation. This is a data collection study in which we ask participants to give us access to information generated before and after RFA treatment of their condition. The RFA procedure uses image guidance to place an electrode through the skin into the target tumor. In RFA, high-frequency electrical currents are passed through an electrode, creating a small region of heat to treat the lesion.

DETAILED DESCRIPTION:
Differentiated thyroid cancer (DTC), which includes papillary and follicular cancer, comprises the vast majority (>90%) of all thyroid cancers. The yearly incidence has nearly tripled from 4.9 per 100,000 in 1975 to 14.3 per 100,000 in 2009. Almost the entire change has been attributed to an increase in the incidence of papillary thyroid cancer (PTC). This increase in incidence is likely driven by the diagnosis of small PTCs <1cm in size due to the increasing use of neck ultrasonography. In a study observing 1235 patients with small papillary thyroid cancer over 22 years, it was noted that at 10 years follow-up, only 8% had tumor enlargement of >3mm and 3.8% had novel lymph node metastases proving that the majority of these 'microcarcinomas' were low-risk and indolent in nature. In 2017, the US commissioned task force evaluating the risks and benefits of treatment of these small cancers concluded that surgical treatment of these microcarcinomas was associated with a low, but not negligible, risk of surgical complications: 2.12-5.93% risk of permanent hypoparathyroidism and 0.99-2.13% risk of permanent recurrent laryngeal nerve injury. In addition, 98.8% of patients treated with thyroidectomy received radioactive iodine that was associated with an excess absolute risk of 11.9 to 13.3 cancers per 10, 000 person-years for second malignancies. In accordance with these data, the most recent societal guidelines for management of thyroid nodules and differentiated thyroid cancer have favored less aggressive management of microcarcinomas, with active surveillance as a reasonable option for management. However, although this may appeal to a subset of individuals who are especially risk and surgery averse, many patients are still uncomfortable with observing 'cancer' and still opt for the least invasive approach to surgical treatment. Thyroid surgery has always been the mainstay of treatment for thyroid cancer. Although associated with excellent outcomes in experienced hands, thyroid surgery carries a low risk of complications that include recurrent or superior laryngeal nerve injury leading to voice changes, hypoparathyroidism, hypothyroidism with need for thyroid hormone supplementation, and unsightly scarring. Although many patients with thyroid cancer find these risks acceptable, these risks are sometimes less acceptable to patients with benign disease. In an era when the medical field is treating thyroid diseases less aggressively, there is a pressing need to identify approaches to treat indolent malignant disease less invasively. Introduced in the early 2000s, ultrasound-guided percutaneous ablation of thyroid lesions has emerged as a potential alternative to surgery in patients with benign thyroid nodules. Of the myriad ablation methods, the most commonly used technique is radiofrequency ablation (RFA). An expanding body of evidence shows that radiofrequency ablation and other percutaneous interventions are effective treatments for benign solid thyroid nodules, toxic adenomas, and thyroid cysts resulting in overall volume reduction ranges of 40-70% with durable resolution of compressive and hyperthyroid symptoms. In addition, RFA has been used as an effective alternative treatment in the management of locally recurrent thyroid cancers in patients who are not good surgical candidates. In addition, RFA of other solid tumors is a commonly performed procedure in the United states and all RFA devices, including the device the investigators will use for the clinical care of these patients, are cleared by the FDA (New devices/technology to the market are approved, but devices that have a predicate device/technology that are already on the market only need to be cleared). Recently, a systematic review and meta-analysis of thermal ablation techniques for micropapillary carcinomas found that among 503 low risk PTCs in 470 patients, no patient experienced tumor recurrence or distant metastasis, 2 patients (0.4%) experienced lymph node metastasis, 1 patient (0.2%) developed a new PTMC, which was successfully treated by additional ablation, and 5 patients (1.1%) underwent delayed surgery after ablation, including the two patients with lymph node metastasis and three additional patients with unknown etiology. Although these percutaneous techniques have been steadily gaining acceptance in Europe and Asia over the past 20 years, they have been slow to be adopted in the US. There remains a dearth of data regarding clinical experience in the United States and no randomized clinical trials have been performed evaluating RFA vs active surveillance for micropapillary carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>/= 18 years)
* Biopsy proven papillary thyroid microcarcinoma (>/= 1.5cm in greatest diameter, PTMC)
* Either refuse surgery or are not good surgical candidates

Exclusion Criteria:

* Cardiac arrhythmia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>/= 18 years) who have a biopsy proven papillary thyroid microcarcinoma (PTMC, >/= 1.5cm in greatest diameter)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Complete sonographic disappearance (CD) | 12 months
  Rate of complete sonographic disappearance of primary tumor s/p RFA

SECONDARY OUTCOMES:
Complications | 12 months
  Procedural complications s/p RFA including but not limited to infection, bleeding, nerve injury, structural injury

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Kuo, MD MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durante C, Costante G, Lucisano G, Bruno R, Meringolo D, Paciaroni A, Puxeddu E, Torlontano M, Tumino S, Attard M, Lamartina L, Nicolucci A, Filetti S. The natural history of benign thyroid nodules. JAMA. 2015 Mar 3;313(9):926-35. doi: 10.1001/jama.2015.0956. PMID 25734734
- [Background] de Rienzo-Madero B, Sabra JP, Gand E, Donatini G, Kraimps JL. Unilateral benign multinodular versus solitary goiter: Long-term contralateral reoperation rates after lobectomy. Surgery. 2019 Jan;165(1):75-79. doi: 10.1016/j.surg.2018.04.074. Epub 2018 Nov 8. PMID 30415868
- [Background] Kim YS, Rhim H, Tae K, Park DW, Kim ST. Radiofrequency ablation of benign cold thyroid nodules: initial clinical experience. Thyroid. 2006 Apr;16(4):361-7. doi: 10.1089/thy.2006.16.361. PMID 16646682
- [Background] Na DG, Lee JH, Jung SL, Kim JH, Sung JY, Shin JH, Kim EK, Lee JH, Kim DW, Park JS, Kim KS, Baek SM, Lee Y, Chong S, Sim JS, Huh JY, Bae JI, Kim KT, Han SY, Bae MY, Kim YS, Baek JH; Korean Society of Thyroid Radiology (KSThR); Korean Society of Radiology. Radiofrequency ablation of benign thyroid nodules and recurrent thyroid cancers: consensus statement and recommendations. Korean J Radiol. 2012 Mar-Apr;13(2):117-25. doi: 10.3348/kjr.2012.13.2.117. Epub 2012 Mar 7. PMID 22438678
- [Background] Kim JH, Baek JH, Lim HK, Ahn HS, Baek SM, Choi YJ, Choi YJ, Chung SR, Ha EJ, Hahn SY, Jung SL, Kim DS, Kim SJ, Kim YK, Lee CY, Lee JH, Lee KH, Lee YH, Park JS, Park H, Shin JH, Suh CH, Sung JY, Sim JS, Youn I, Choi M, Na DG; Guideline Committee for the Korean Society of Thyroid Radiology (KSThR) and Korean Society of Radiology. 2017 Thyroid Radiofrequency Ablation Guideline: Korean Society of Thyroid Radiology. Korean J Radiol. 2018 Jul-Aug;19(4):632-655. doi: 10.3348/kjr.2018.19.4.632. Epub 2018 Jun 14. PMID 29962870
- [Background] Gharib H, Papini E, Garber JR, Duick DS, Harrell RM, Hegedus L, Paschke R, Valcavi R, Vitti P; AACE/ACE/AME Task Force on Thyroid Nodules. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS, AMERICAN COLLEGE OF ENDOCRINOLOGY, AND ASSOCIAZIONE MEDICI ENDOCRINOLOGI MEDICAL GUIDELINES FOR CLINICAL PRACTICE FOR THE DIAGNOSIS AND MANAGEMENT OF THYROID NODULES--2016 UPDATE. Endocr Pract. 2016 May;22(5):622-39. doi: 10.4158/EP161208.GL. PMID 27167915
- [Background] Jeong WK, Baek JH, Rhim H, Kim YS, Kwak MS, Jeong HJ, Lee D. Radiofrequency ablation of benign thyroid nodules: safety and imaging follow-up in 236 patients. Eur Radiol. 2008 Jun;18(6):1244-50. doi: 10.1007/s00330-008-0880-6. Epub 2008 Feb 20. PMID 18286289
- [Background] Baek JH, Kim YS, Lee D, Huh JY, Lee JH. Benign predominantly solid thyroid nodules: prospective study of efficacy of sonographically guided radiofrequency ablation versus control condition. AJR Am J Roentgenol. 2010 Apr;194(4):1137-42. doi: 10.2214/AJR.09.3372. PMID 20308523
- [Background] Watt T, Barbesino G, Bjorner JB, Bonnema SJ, Bukvic B, Drummond R, Groenvold M, Hegedus L, Kantzer V, Lasch KE, Marcocci C, Mishra A, Netea-Maier R, Ekker M, Paunovic I, Quinn TJ, Rasmussen AK, Russell A, Sabaretnam M, Smit J, Torring O, Zivaljevic V, Feldt-Rasmussen U. Cross-cultural validity of the thyroid-specific quality-of-life patient-reported outcome measure, ThyPRO. Qual Life Res. 2015 Mar;24(3):769-80. doi: 10.1007/s11136-014-0798-1. Epub 2014 Sep 7. PMID 25194574
- [Background] Dobnig H, Amrein K. Monopolar Radiofrequency Ablation of Thyroid Nodules: A Prospective Austrian Single-Center Study. Thyroid. 2018 Apr;28(4):472-480. doi: 10.1089/thy.2017.0547. Epub 2018 Mar 20. PMID 29490593